CLINICAL TRIAL: NCT01758276
Title: Obstetric Complications in Women Who Smoke During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0092-12
Record Dates: First submitted 2012-12-26; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: Smoking
Keywords: smoking, pregnancy
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non smokers: Women who did not report smoking in pregnancy
- Smokers in pregnancy: Women who report smoking in pregnancy

SUMMARY:
This will be a retrospective study. Details on all women who delivered in McGill University between 2001-2007 will be retrieved anonymously from the MOND database (McGill University Obstetrics and Neonatal database). Women will be divided to 2 groups according to their smoking status in pregnancy. Obstetric complications will be recorded in both groups.

DETAILED DESCRIPTION:
This will be a retrospective study using the McGill University Obstetrics and Neonatal database (MOND). This is a comprehensive database the contains details on all women delivering in McGill University Health Center in Montreal Canada.

Details on all women who delivered in McGill University between 2001-2007 will be retrieved anonymously from the MOND database (McGill University Obstetrics and Neonatal database). Women will be divided to 2 groups according to their smoking status in pregnancy. Obstetric complications will be recorded in both groups.

Statistic tests would be applied in order to assess relation between smoking and Obstetrical complications.

ELIGIBILITY:
Inclusion Criteria:all

* All women who delivered in McGill University health center between 2001-2008

Exclusion Criteria:

* delivery prior to 24 weeks (data on <24 weeks not included in the database..)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women who delivered in McGill University health center between 2001-2008
Sampling Method: Probability Sample
Enrollment: 21000 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal Intensive Care Unit admission rate in women who smoke in pregnancy | pregnancy 40 weeks
  Using the MOND database We will assess NICU admission rate of babies to women who smoke

SECONDARY OUTCOMES:
Birthweight | 40 weeks of pregnancy
  we will assess birth weight of babies to mothers who smoke Vs those who don't

CONTACTS AND LOCATIONS:
Overall Officials: Alon Shrim, MD, Principal Investigator — Hillel Yaffe Medical Center